CLINICAL TRIAL: NCT05941962
Title: Use of Hand-held Dynamometry to Obtain Objective Measures of Lower Extremity Rate of Peak Force Production, Cumulative Peak Force Production, and Sustained Peak Force Production Among Patients With Chronic Stroke
Brief Title: Use of Hand-held Dynamometry to Obtain Objective Measures of Lower Extremity Force Production With Chronic Stroke
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Cathey Norton, Primary Investigator, Vanderbilt University Medical Center
Other Study IDs: 230030
Record Dates: First submitted 2023-06-05; First posted 2023-07-12 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-05

CONDITIONS: Chronic Stroke; Weakness, Muscle
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Average Force Production: Average force production of bilateral lower extremities will be collected using the handheld dynamometer, Activbody Activ5.

SUMMARY:
This study wants to know if using handheld dynamometry (HHD) to test leg strength in persons who have had a stroke, will reduce mistakes and give therapists better information to use for therapy. This study will collect normal values of leg muscle peak force production, cumulative peak force production, and sustained peak force production in patients with chronic stroke.

DETAILED DESCRIPTION:
The Activbody Activ5 device will be used for data collection with all information logged and stored through the device's app and transferred to secure files. Assessment of isometric muscle strength and power will be performed as follows:

* Hip flexors with the participant seated and hips and knees flexed at 90 degrees
* Knee extensors with the participant seated and hips and knees flexed at 90 degrees
* Knee flexors with the participant seated and hips and knees flexed at 90 degrees
* Ankle plantarflexors with the participant lying supine with the ankle in plantargrade and hips and knees extended
* Ankle dorsiflexors with the participant lying supine with the ankle relaxed and hips and knees extended
* Hip abductors with the participant lying supine and hips and knees extended
* Hip adductors with the participant lying supine and hips and knees extended
* Hip extensors with the participant lying prone and hips and knees extended 1 session, two trials per side

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Stroke > 3 months
* Ability to follow two-step commands
* Ability to assume all test positions and maintain for duration of testing (i.e. upright seated, prone, side lying, supine)

Exclusion Criteria:

* Lower extremity contractures preventing full passive range of motion (ROM)
* Vital signs contraindicated for exercise (i.e. resting heart rate > 100 bpm < 50 bpm, resting systolic blood pressure > 200 mmHg or < 90 mmHg, resting diastolic blood pressure > 110 mmHg, oxygen saturation < 90%)
* Symptoms contraindicated for testing (i.e. shortness of breath, angina, dizziness, severe headache, sudden onset of numbness or weakness, painful calf suggestive of deep vein thrombosis)
* Active infection and/or injury at location of testing site
* Other diagnosed co-morbidities that would impact physical participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Age 18 years or older
  - Stroke > 3 months
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2025-07-26 (Actual); Study Completion 2025-07-26 (Actual)

PRIMARY OUTCOMES:
Hand-held Dynamometry Measurement of Average Force Production | 1 year
  Average force production of lower extremity isometric strength measured in pounds (lb)

SECONDARY OUTCOMES:
Hand-held Dynamometry Measurement of Peak Force Production | 1 year
  Peak force production of lower extremity isometric strength measured in pounds (lb)

OTHER OUTCOMES:
Hand-held Dynamometry Measurement of Time to Peak Force | 1 year
  Time required to reach peak force production of lower extremity isometric strength measured in seconds (sec)

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Andrews AW, Bohannon RW. Short-term recovery of limb muscle strength after acute stroke. Arch Phys Med Rehabil. 2003 Jan;84(1):125-30. doi: 10.1053/apmr.2003.50003. PMID 12589633
- [Result] Bakers JNE, van den Berg LH, Ajeks TG, Holleman MJ, Verhoeven J, Beelen A, Visser-Meily JMA, van Eijk RPA. Portable fixed dynamometry: towards remote muscle strength measurements in patients with motor neuron disease. J Neurol. 2021 May;268(5):1738-1746. doi: 10.1007/s00415-020-10366-9. Epub 2020 Dec 23. PMID 33355879
- [Result] Bohannon RW. Considerations and Practical Options for Measuring Muscle Strength: A Narrative Review. Biomed Res Int. 2019 Jan 17;2019:8194537. doi: 10.1155/2019/8194537. eCollection 2019. PMID 30792998
- [Result] Mentiplay BF, Perraton LG, Bower KJ, Adair B, Pua YH, Williams GP, McGaw R, Clark RA. Assessment of Lower Limb Muscle Strength and Power Using Hand-Held and Fixed Dynamometry: A Reliability and Validity Study. PLoS One. 2015 Oct 28;10(10):e0140822. doi: 10.1371/journal.pone.0140822. eCollection 2015. PMID 26509265
- [Result] Mentiplay BF, Tan D, Williams G, Adair B, Pua YH, Bower KJ, Clark RA. Assessment of isometric muscle strength and rate of torque development with hand-held dynamometry: Test-retest reliability and relationship with gait velocity after stroke. J Biomech. 2018 Jun 25;75:171-175. doi: 10.1016/j.jbiomech.2018.04.032. Epub 2018 Apr 27. PMID 29731325
- [Result] Merry K, Napier C, Chung V, Hannigan BC, MacPherson M, Menon C, Scott A. The Validity and Reliability of Two Commercially Available Load Sensors for Clinical Strength Assessment. Sensors (Basel). 2021 Dec 16;21(24):8399. doi: 10.3390/s21248399. PMID 34960492
- [Result] Shefner JM. Strength Testing in Motor Neuron Diseases. Neurotherapeutics. 2017 Jan;14(1):154-160. doi: 10.1007/s13311-016-0472-0. PMID 27600518
- See also: Short-term recovery of limb muscle strength after acute stroke. Archives of Physical Medicine and Rehabilitation — https://doi.org/10.1053/apmr.2003.50003
- See also: Portable fixed dynamometry: Towards remote muscle strength measurements in patients with motor neuron disease. — https://doi.org/10.1007/s00415-020-10366-9
- See also: Assessment of lower limb muscle strength and power using hand-held and fixed dynamometry: A reliability and validity study. — https://doi.org/10.1371/journal.pone.0140822
- See also: Assessment of isometric muscle strength and rate of torque development with hand-held dynamometry: Test-retest reliability and relationship with gait velocity after stroke. — https://doi.org/10.1016/j.jbiomech.2018.04.032
- See also: Strength testing in motor neuron diseases. — https://doi.org/10.1007/s13311-016-0472-0